CLINICAL TRIAL: NCT05001750
Title: Are Long Term Prophylactic Antibiotics Useful With Antibiotic Impregnated External Ventricular Drains (EVDs)?
Brief Title: Prophylactic Antibiotics Useful With Antibiotic Impregnated External Ventricular Drains (EVDs)?
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12680
Record Dates: First submitted 2021-06-25; First posted 2021-08-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Subarachnoid Hemorrhage; Intracerebral Hemorrhage; Ventriculitis, Cerebral; Hydrocephalus
Keywords: Subarachnoid hemorrhage; Intracerebral Hemorrhage; Ventriculitis; Hydrocephalus
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebral Hemorrhage; Cerebral Ventriculitis; Hydrocephalus | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into one of two groups, either continuous antibiotic usage until the EVD is removed or antibiotics for a total of twenty-four hours; in both cases antibiotics will begin no more than sixty minutes pre-procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continuous antibiotic use until the EVD is removed (Experimental): Continuous prophylactic antibiotic use until the EVD is removed. Antibiotics will begin no more than sixty minutes pre-procedure.
  Interventions: Drug: Long term (continuous) prophylactic antibiotics
- Antibiotics for a total of twenty-four hours (Experimental): Antibiotics for a total of twenty-four hours. Antibiotics will begin no more than sixty minutes pre-procedure.
  Interventions: Drug: 24 hours antibiotics

INTERVENTIONS:
Drug: Long term (continuous) prophylactic antibiotics — VRIs in patients who also receive a pre-procedural dose of antibiotics with continued dosing of antibiotics for the duration of the external ventricular drain. Nafcillin 1-2 grams every 6 hours (depending on weight) until the EVD is removed. If penicillin allergic, Doxycycline 100mg every 12 hours until the EVD is removed.
  Arms: Continuous antibiotic use until the EVD is removed
Drug: 24 hours antibiotics — Nafcillin 1-2 grams every 6 hours (depending on weight) for a total of 24 hours. If penicillin allergic, Doxycycline 100mg every 12 hours for a total of 24 hours.
  Arms: Antibiotics for a total of twenty-four hours

SUMMARY:
The principal objective of this study is to compare the incidence of ventriculostomy related infections (VRIs) in patients who receive twenty-four hours of antibiotics, beginning no more than sixty minutes prior to EVD placement, to the incidence of VRIs in patients who also receive a pre-procedural dose of antibiotics with continued dosing of antibiotics for the duration of the external ventricular drain (EVD). At this time, the duration of prophylactic antibiotic use with antibiotic impregnated EVDs is unknown.

DETAILED DESCRIPTION:
Intracranial hemorrhage (ICH), which include subarachnoid hemorrhage (SAH), intraparenchymal hemorrhage (IPH) and intraventricular hemorrhage (IVH) affects nearly 30,000 every year in US alone. Despite rapid advances in treatment of just one of these pathologies, SAH, the case fatality rate remains at 32.2% in US. Successful post interventional outcome of patients suffering from SAH depends on the management of a multitude of secondary neurological complications, including prevention of re-hemorrhage, vasospasm, hydrocephalus, increased intracranial pressure (ICP), and seizure. A major component of this care is placement of an external ventricular drain (EVD), which is routine in patients suffering from SAH to manage ICP and to treat hydrocephalus.

Placement of an EVD, however, is not without risk, in particular with regards to infection, commonly referred to as Ventriculostomy Related Infection (VRI). The rate of VRIs has been reported to range widely from 0% to 40% however, with an increased risk in patients suffering from hemorrhage or any vascular diseases (28.6%) in this subgroup, while typically lower (18.5%) in patients suffering from other neurosurgical diagnoses.

Ventriculostomy related infections have been associated with increased delayed cerebral ischemia (a.k.a.; vasospasm), extended hospital duration, increased mortality and higher hospital costs. Despite the importance of management and prevention of VRIs, there hasn't been any clear consensus on administration of antibiotics post-procedurally. This is perpetuated by the fact that each institution, and even providers within institutions, have varying definitions of VRIs, and their own protocols regarding administration of antibiotics.

Although there is an established protocol for insertion of EVD, which include pre-procedural intravenous antibiotic administration, there is no consensus on duration of post-operative antibiotics, despite the fact that successful patient outcomes depend on management of these VRIs.

Further complicating the problem is the growing concern over increasing resistance to gram-positive organisms due to overuse of systemic antibiotics, as well as development of Clostridium difficile infection. As a result, practice is quite variable, based upon individual clinician preferences, rather than evidence based. Determining optimal strategies and protocols to minimize the incidence of VRI, while ensuring responsible antibiotic usage, thereby minimizing their deleterious effects on both individuals and communities, is of chief interest.

These universal concerns and questions deserve a new formal study in this initial feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18 years
* patients diagnosed with a subarachnoid hemorrhage, intracerebral hemorrhage, or acute ischemic stroke who require an EVD for management of their underlying condition. In certain cases (a small minority), an EVD must be replaced due to failure (i.e., blood clot interrupting flow). In such cases, patients will be re-dosed with antibiotics prior to catheter exchange in typical fashion and continue in their previously randomized treatment group

Exclusion Criteria:

* patients who were on antibiotics within the week prior to admission
* patients with leukopenia (<5000) at baseline
* patients with signs of meningitis, ventriculitis or any other infection at presentation
* patients who are pregnant or prisoners
* patients aged < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Cerebrospinal Fluid Positive (CSF+) VRI | From EVD insertion until discharge - estimated period of time is 2 weeks
  A VRI will be defined as an infection of the CNS including abscess (when occurring after EVD placement), ventriculitis, or meningitis. To receive a diagnosis of meningitis or ventriculitis, NHSN criteria (1) OR (2) must be met:
  1. Patient has organism(s) identified from CSF by a culture or non-culture based microbiological method (PCR) performed for purposes of clinical diagnosis or treatment
     OR
  2. Patient has 2 or more of:
     1. fever (>38.0°C) or headache
     2. meningeal sign(s)
     3. cranial nerve sign(s)
        AND 1 or more of:
     4. increased white cells, elevated protein, and decreased glucose in CSF (per reporting lab's reference range)
     5. organism(s) seen on Gram stain of CSF
     6. organism(s) identified from blood by a culture or non-culture based microbiologic testing method performed for purposes of clinical diagnosis or treatment (not Active Surveillance Culture/Testing)
     7. diagnostic single antibody titer (IgM) or 4-fold increase in paired sera (IgG) for organism

SECONDARY OUTCOMES:
Class of infecting organism | From EVD insertion until discharge - estimated period of time is 2 weeks
  Class of infecting organisms identified will be summarized by study arm to assess whether the infections that occur in both treatment groups are caused by the same type of pathogen. The class of infecting organism will be summarized by study arm.
Time to infection | From EVD insertion until discharge - estimated period of time is 2 weeks
  Time to infection will be assessed from the time of EVD placement until discharge. Results will be summarized by study arm using descriptive statistics.
Number of attempts at EVD catheter insertion | From EVD insertion until discharge - estimated period of time is 2 weeks
  The number of attempts to insert the catheter will be evaluated. This outcome will be used to determine any subsequent effect catheter placement may have had on incidence of infection for each treatment modality. The number of placement attempts will be summarized by study arm.
Incidence of nosocomial infections | From EVD insertion until discharge - estimated period of time is 2 weeks
  The incidence of nosocomial infections of C. difficile or other multidrug resistant nosocomial infections in participants will be evaluated. Incidence in the context of this study will equal the number of new EVD-related infections divided by the total EVD days at risk and expressed as a percentage. Results will be summarized by study arm using descriptive statistics.
Overall Morbidity | From EVD insertion until discharge - estimated period of time is 2 weeks
  Overall morbidity, defined as morbidity from all causes, will be determined. This will include any morbidity from high grade fever (>101 degrees Fahrenheit), repositioning of EVD, post procedural hemorrhage, or new catheter placement due to new bleeding (at a different location than original), or need for permanent CSF drainage (i.e. ventriculoperitoneal shunt). Morbidity will be summarized by study arm.
Overall Mortality | From EVD insertion until discharge - estimated period of time is 2 weeks
  Overall mortality, defined as mortality from all causes, will be determined. Mortality along with cause of death will be recorded and summarized for patients who die during the period of insertion of EVD until one week after its removal.

CONTACTS AND LOCATIONS:
Overall Officials: David C Altschul, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nieuwkamp DJ, Setz LE, Algra A, Linn FH, de Rooij NK, Rinkel GJ. Changes in case fatality of aneurysmal subarachnoid haemorrhage over time, according to age, sex, and region: a meta-analysis. Lancet Neurol. 2009 Jul;8(7):635-42. doi: 10.1016/S1474-4422(09)70126-7. Epub 2009 Jun 6. PMID 19501022
- [Background] Lozier AP, Sciacca RR, Romagnoli MF, Connolly ES Jr. Ventriculostomy-related infections: a critical review of the literature. Neurosurgery. 2002 Jul;51(1):170-81; discussion 181-2. doi: 10.1097/00006123-200207000-00024. PMID 12182415
- [Background] Foreman PM, Chua M, Harrigan MR, Fisher WS 3rd, Vyas NA, Lipsky RH, Walters BC, Tubbs RS, Shoja MM, Griessenauer CJ. Association of nosocomial infections with delayed cerebral ischemia in aneurysmal subarachnoid hemorrhage. J Neurosurg. 2016 Dec;125(6):1383-1389. doi: 10.3171/2015.10.JNS151959. Epub 2016 Feb 12. PMID 26871202
- [Background] Frontera JA, Fernandez A, Schmidt JM, Claassen J, Wartenberg KE, Badjatia N, Parra A, Connolly ES, Mayer SA. Impact of nosocomial infectious complications after subarachnoid hemorrhage. Neurosurgery. 2008 Jan;62(1):80-7; discussion 87. doi: 10.1227/01.NEU.0000311064.18368.EA. PMID 18300894
- [Background] Lyke KE, Obasanjo OO, Williams MA, O'Brien M, Chotani R, Perl TM. Ventriculitis complicating use of intraventricular catheters in adult neurosurgical patients. Clin Infect Dis. 2001 Dec 15;33(12):2028-33. doi: 10.1086/324492. Epub 2001 Nov 9. PMID 11712094
- [Background] Aucoin PJ, Kotilainen HR, Gantz NM, Davidson R, Kellogg P, Stone B. Intracranial pressure monitors. Epidemiologic study of risk factors and infections. Am J Med. 1986 Mar;80(3):369-76. doi: 10.1016/0002-9343(86)90708-4. PMID 3953614
- [Background] Mayhall CG, Archer NH, Lamb VA, Spadora AC, Baggett JW, Ward JD, Narayan RK. Ventriculostomy-related infections. A prospective epidemiologic study. N Engl J Med. 1984 Mar 1;310(9):553-9. doi: 10.1056/NEJM198403013100903. PMID 6694707
- [Background] Wong GK, Poon WW. Ventriculostomy infections. J Neurosurg. 2006 Sep;105(3):506-7; author reply 507. doi: 10.3171/jns.2006.105.3.506. No abstract available. PMID 16961156
- [Background] Poblete R, Zheng L, Raghavan R, Cen S, Amar A, Sanossian N, Mack W, Kim-Tenser M. Trends in Ventriculostomy-Associated Infections and Mortality in Aneurysmal Subarachnoid Hemorrhage: Data From the Nationwide Inpatient Sample. World Neurosurg. 2017 Mar;99:599-604. doi: 10.1016/j.wneu.2016.12.073. Epub 2016 Dec 27. PMID 28034809
- [Background] Camacho EF, Boszczowski I, Basso M, Jeng BC, Freire MP, Guimaraes T, Teixeira MJ, Costa SF. Infection rate and risk factors associated with infections related to external ventricular drain. Infection. 2011 Feb;39(1):47-51. doi: 10.1007/s15010-010-0073-5. Epub 2011 Jan 25. PMID 21264679